CLINICAL TRIAL: NCT05597722
Title: Randomized Study to Evaluate Strategies to Address Cognitive Fog in Long-COVID-19 Patients
Brief Title: Addressing Cognitive Fog in Long-COVID-19 Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the evolving nature of COVID-related cognitive fog, it was determined that the study would be terminated at this time. The team agreed that it isn't feasible to collect enough data to evaluate the efficacy of the treatments.
Sponsor: Eva Szigethy (Other)
Collaborators: The Beckwith Institute (Other)
Responsible Party: Sponsor-Investigator, Eva Szigethy, Professor of Psychiatry Pediatrics and Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22050191
Record Dates: First submitted 2022-10-27; First posted 2022-10-28 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Impairment; Long COVID
Keywords: Cognitive fog, Long-COVID
MeSH Terms: conditions — Cognitive Dysfunction; Post-Acute COVID-19 Syndrome | interventions — SLI381; Adderall

STUDY DESIGN:
Intervention Model Description: This is a randomized 1:1 block design trial evaluating the effect of a digital cognitive behavioral app versus a drug therapy (amphetamine-dextroamphetamine [Adderall]) on cognitive impairment and other secondary outcomes in subjects with post-COVID symptoms (Long-COVID). The participants will be stratified by depression severity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital cognitive behavioral intervention- RxWell (Active Comparator): The mobile app provides users with brief skill building techniques such as relaxation, behavioral activation and exposure, distress tolerance, cognitive reframing, and mindfulness meditation, for anxiety and depression. The content of RxWell was developed based on standard CBT techniques for treating anxiety disorders and depression. The user will have the option to select either the depression or anxiety program, and the coach will have the ability to personalize the program so that the individual can utilize the proper CBT techniques that fits with their presentation.
  The health coach communicates with RxWell users via asynchronous, secure within app messaging. They reinforce CBT principles, guide users through goal setting, and help users work through challenges and recognize successes. The coaches will also receive individualized cognitive rehabilitation tips from the speech therapist after their appointment with the participant.
  Interventions: Behavioral: Digital cognitive behavioral intervention-RxWell
- Stimulant Medication (Active Comparator): The other intervention is a stimulant medication known to reduce cognitive impairment in other chronic medical conditions, such as Inflammatory Bowel Disease. The Long-COVID psychiatrist will order the medication and the participant will be scheduled for a 6-week research tele visit with the psychiatrist to monitor for any medication side effects. Amphetamine-dextroamphetamine drug dose will be 10mg daily for 12 weeks, and no dose changes will be made. Amphetamine-dextroamphetamine is a Schedule II controlled substance that has a risk for abuse, tolerance, and psychological dependence, which can be associated with severe social disability.
  Interventions: Drug: Amphetamine-Dextroamphetamine

INTERVENTIONS:
Behavioral: Digital cognitive behavioral intervention-RxWell — RxWell is a coach enhanced digital behavioral health intervention that teaches techniques to help manage emotional distress, which may improve cognitive fog and/or depression. Participants will have access to this app for three months.
  Arms: Digital cognitive behavioral intervention- RxWell
Drug: Amphetamine-Dextroamphetamine — Participants randomized to this arm will be prescribed 10mg of amphetamine-dextroamphetamine to take as needed to help with cognitive fog. Participants in this arm will be contacted at 2 and 6 weeks to assess for any side effects from taking the medication.
  Other Names: Adderall
  Arms: Stimulant Medication

SUMMARY:
This study will assess two options to help patients better manage the cognitive fog and emotional distress that may be associated with having Long-COVID. Long-COVID is post-COVID conditions or symptoms lasting more than four weeks after infection. Clinicians from the UPMC Long-COVID Clinic leading this study are evaluating the utility of computer-based evaluation of COVID-related cognitive fog and the helpfulness of two intervention strategies to treat moderate cognitive impairment using a randomized trial. The two intervention strategies include 1) a standardized dosing of amphetamine/dextroamphetamine medication that has been used to improve cognitive fog; and 2) a digital behavioral tool with an embedded health coach that is used on a mobile phone.

DETAILED DESCRIPTION:
Eligible participants will be randomized to one of two arms. One intervention targets cognitive fog associated with depression (RxWell mobile app), the other the cognitive fog directly (Amphetamine-dextroamphetamine medication). Two weeks after randomization, participants are contacted by study staff to complete the GAD7. Participants who are randomized to RxWell will be offered assistance if they were not able to download the app on their own. Participants who are randomized to receive the stimulant will also complete a stimulant drug side effect rating scale to determine if the participant has any effects from the medication.

All participants will complete computerized neurocognitive assessments (ImPACT, and BrainCheck) and other study measures (MOCA (Screen, 1.5 and 3 months), Patient Health Questionnaire, Generalized Anxiety Disorder Measure, Satisfaction with Life Scale, PCL-5 Post Traumatic Stress Disorder checklist, ADHD Symptom Screener, and Sheehan Disability Scale) at baseline, 1.5 (interim) and 3 months after randomization. The study measures, other than the neuro-cognitive assessments, will be completed via REDCap.

ELIGIBILITY:
Inclusion Criteria:

* History of SARS-CoV-2 infection as defined as a positive PCR or home antigen test
* Patients with Long-COVID as defined as COVID symptoms that persist for three months or longer.
* Between the ages of 21 and 65
* Moderate cognitive impairment (MOCA score to meet criteria is < or =18) present for at least 3 months
* Response of "No" to the screening question, "Are you pregnant or do you plan to become pregnant in the next 3 months?"
* Access to a smartphone

Exclusion Criteria:

* History of dementia, psychosis, mania, addiction or current conditions requiring immediate hospitalization
* Previous adverse or allergic reaction to Adderall or other amphetamines
* Pre-existing cardiac or kidney condition, severe hypertension, glaucoma, advanced arteriosclerosis, hyperthyroidism, and taking an MAOI within the past 14 days
* Current or past substance misuse
* Previous use of RxWell (completed 3 or more techniques)
* Current use of amphetamine-dextroamphetamine
* History of uncontrolled blood pressure
* Subjects taking Methylphenidate; Lisdexamfetamine; non-Adderall amphetamine products; Atomoxetine; Viloxazine; Modafinil; Armodafinil; Nortriptyline and other tricyclic drugs; Bupropion; Tramadol; and Monoamine Oxidase Inhibitor (MAOI) drugs (including Linezolid).
* Inability to pay for study medication.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Data is shared at the aggregate level.

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Cognitive Behavioral Intervention- RxWell: The mobile app provides users with brief skill building techniques such as relaxation, behavioral activation and exposure, distress tolerance, cognitive reframing, and mindfulness meditation, for anxiety and depression. The content of RxWell was developed based on standard CBT techniques for treating anxiety disorders and depression. The user will have the option to select either the depression or anxiety program, and the coach will have the ability to personalize the program so that the individual can utilize the proper CBT techniques that fits with their presentation.
  The health coach communicates with RxWell users via asynchronous, secure within app messaging. They reinforce CBT principles, guide users through goal setting, and help users work through challenges and recognize successes. The coaches will also receive individualized cognitive rehabilitation tips from the speech therapist after their appointment with the participant.
  Digital cognitive behavioral intervention-RxWell: RxWell is a coach enhanced digital behavioral health intervention that teaches techniques to help manage emotional distress, which may improve cognitive fog and/or depression. Participants will have access to this app for three months.
Period: Overall Study
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Started | 6 | 1
Completed | 0 | 0
Not Completed | 6 | 1
Not completed — Study was terminated | 6 | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated prior to any baseline assessments being analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41 [27 to 60] | 47 [47 to 47] | 42 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Impairment - MOCA
Description: The MOCA is a validated screening tool that provides a total score to assess for mild cognitive impairment.
Time Frame: Compare baseline to 12 weeks
Population: The trial was terminated before the outcome measure data were collected. No follow-up data was collected for any participant.
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Cognitive Impairment - BrainCheck
Description: BrainCheck is an FDA approved validated, automated, remote neurocognitive assessments in multiple domains.
Time Frame: Compare baseline to 12 weeks
Population: as for outcome 1
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Cognitive Impairment - ImPACT
Description: ImPACT is an FDA approved computerized neurocognitive concussion assessment tool that provides composite sores to evaluate cognitive abilities.
Time Frame: Compare baseline to 12 weeks
Population: as for outcome 1
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Depression - PHQ8
Description: Patient Health Questionnaire (PHQ8) will be utilized to measure change in depression severity from baseline up to 12 weeks after baseline.
  The PHQ-8 is an 8 item questionnaire. Scores can range from 0-24. A score of 0-4 indicates no depressive symptoms; 5-9 indicates mild depressive symptoms; 10-19 indicates moderate depressive symptoms; 20-24 indicates severe depressive symptoms.
Time Frame: Compare baseline up to 12 weeks
Population: as for outcome 1
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Quality of Life - SWLS
Description: Satisfaction with Life Scale (SWLS) will be utilized to measure change in quality of life from baseline up to 12 weeks after baseline.
  SWLS is a five item measure with a maximum score of 35. Higher score correlate with higher satisfaction of life. Scores 31-35 extremely satisfied. Scores less than 9 indicate extremely dissatisfied.
Time Frame: Compare baseline up to 12 weeks
Population: as for outcome 1
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Disability
Description: Sheehan Disability Scale assess functional impairment in three inter-related domains; work/school, social and family life. The three items are summed into a single measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Compare baseline up to 12 weeks
Population: as for outcome 1
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the one month participants were involved in the study prior to the termination of the study.
Description: The 1 subject randomized to the stimulant arm never received the medication. 2 of the 6 subjects randomized to RxWell downloaded the app.
Arm/Group | Digital Cognitive Behavioral Intervention- RxWell | Stimulant Medication
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05597722/Prot_SAP_000.pdf